CLINICAL TRIAL: NCT01942733
Title: Interventional, Open-label, Flexible-dose, Exploratory Study of Brexpiprazole as Adjunctive Treatment of Sleep Disturbances in Patients With Major Depressive Disorder
Brief Title: Study of Brexpiprazole as Adjunctive Treatment of Sleep Disturbances in Patients With Major Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15352A
Record Dates: First submitted 2013-09-11; First posted 2013-09-16 (Estimated); Results first posted 2016-03-01 (Estimated); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Sleep Disturbances
MeSH Terms: conditions — Parasomnias | interventions — brexpiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Brexpiprazole (Experimental): Brexpiprazole adjunct to open-label treatment with a commercially available antidepressant treatment (ADT)
  Interventions: Drug: Brexpiprazole

INTERVENTIONS:
Drug: Brexpiprazole — 2-3 mg/day, once daily, tablets, for oral use. The patients received 1mg/day brexpiprazole during Week 1 and 2mg/day during Week 2 (up-titration) and from Weeks 3 to 6 they received 3mg/day; depending on tolerability the dose could be reduced to 2mg/day based on the investigator's judgment.

SUMMARY:
To assess effects of brexpiprazole on sleep patterns of depressed patients with sleep disturbances.

ELIGIBILITY:
Inclusion Criteria - at Screening:

* The patient has a Major Depressive Episode (MDE) associated to Major Depressive Disorder (MDD), diagnosed according to Diagnostic and Statistical Manual of Mental Disorders, 4th edition, Text Revision (DSM-IV-TR™). The current MDE should be confirmed using the Mini International Neuropsychiatric Interview (MINI).
* The patient has an inadequate response to at least one antidepressant treatment (including the treatment the patient is taking at screening) in the current MDE, as documented by self-report as less than a pre-defined response on the Massachusetts General Hospital Antidepressant Treatment Response Questionnaire (ATRQ).
* The patient has a pre-defined Montgomery Aasberg Depression Rating Scale (MADRS) total score, and a pre-defined Clinical Global Impression - Severity of Illness (CGI-S) score at screening, and has had the current MDE for ≥10 weeks.
* The patient is currently treated for the current MDE with an adequate selective serotonin reuptake inhibitor (SSRI) or a serotonin-norepinephrine reuptake inhibitor (SNRI) antidepressant treatment for ≥6 weeks, at the same dosage for ≥2 weeks.
* The patient has sleep disturbances (difficulty falling asleep and/or difficulty staying asleep and/or problem waking up too early) confirmed by a pre-defined Insomnia Severity Index (ISI) score.
* The patient agrees to protocol-defined use of effective contraception.

Entry Criteria to Treatment Period (Baseline Visit):

* The patient still fulfils DSM-IV-TR™ criteria for MDE.
* The patient received the same SSRI or SNRI antidepressant treatment at adequate dose during the entire lead-in period.
* The patient has a pre-defined MADRS total score.
* The patient's improvement in the MADRS total score is a pre-defined percentage compared to screening.
* The patient has a pre-defined Clinical Global Impression - Global Improvement (CGI-I) score.
* The patient has sleep disturbances (difficulty falling asleep and/or difficulty staying asleep and/or problem waking up too early) confirmed by a pre-defined ISI score.
* The patient has sleep disturbances confirmed by pre-defined Latency to Persistent Sleep (LPS) and pre-defined Sleep Efficiency (SE).

Exclusion Criteria:

- The patient is, in the investigator's opinion, unlikely to comply with the protocol or is unsuitable for any reason.

Other inclusion and exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2013-09; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com

REFERENCES:
- [Derived] Krystal AD, Mittoux A, Lindsten A, Baker RA. Chronobiologic parameter changes in patients with major depressive disorder and sleep disturbance treated with adjunctive brexpiprazole: An open-label, flexible-dose, exploratory substudy. J Affect Disord. 2021 Jan 1;278:288-295. doi: 10.1016/j.jad.2020.09.026. Epub 2020 Sep 11. PMID 32979560
- [Derived] Krystal AD, Mittoux A, Meisels P, Baker RA. Effects of Adjunctive Brexpiprazole on Sleep Disturbances in Patients With Major Depressive Disorder: An Open-Label, Flexible-Dose, Exploratory Study. Prim Care Companion CNS Disord. 2016 Sep 8;18(5). doi: 10.4088/PCC.15m01914. PMID 27835722

RESULTS

PARTICIPANT FLOW:
Groups:
- Brexpiprazole: Brexpiprazole adjunct to open-label treatment with a commercially available antidepressant treatment (ADT)
  Brexpiprazole: 2-3 mg/day, once daily, tablets, for oral use
Period: Overall Study
Arm/Group | Brexpiprazole
Started | 44
Completed | 41
Not Completed | 3
Not completed — Lost to Follow-up | 1
Not completed — Non-compliance with IMP | 1
Not completed — Administrative | 1

BASELINE CHARACTERISTICS:
Population: The all-patients-treated set (APTS) comprises all patients who took at least one dose of brexpiprazole.
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.4 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 16
  White | 24
  More than one race | 0
  Unknown or Not Reported | 1
MADRS total score [Mean (Standard Deviation); unit: units on a scale] — The Montgomery and Åsberg Depression Rating Scale (MADRS) is a 10-item rating scale designed to assess the severity of the symptoms in depressive illness and to be sensitive to treatment effects. Symptoms are rated on a 7-point scale from 0 (no symptom) to 6 (severe symptom). The total score of the 10 items ranges from 0 to 60, with higher values indicating worse outcome. The overall number of baseline participants was based on the full analysis set (FAS)(n=54).
  units on a scale | 28.3 (3.8)
CGI-S score [Mean (Standard Deviation); unit: units on a scale] — The Clinical Global Impression - Severity of Illness (CGI-S) scale assesses the clinician's impression of the patient's current state of mental illness. The clinician uses his or her clinical experience of this patient population to rate the severity of the patient's current mental illness on a 7-point scale ranging from 1 (normal - not at all ill) to 7 (among the most extremely ill patients), with higher values indicating worse outcome. The overall number of baseline participants was based on the full analysis set (FAS)(n=44).
  units on a scale | 4.3 (0.8)
ESS total score [Mean (Standard Deviation); unit: units on a scale] — The Epworth Sleepiness Scale (ESS) is a is a patient-rated scale designed to measure daytime sleepiness. The ESS consists of 8 items describing different situations/activities and the patients rate the chance of them dozing off or falling asleep when they are in these situations. Each item is rated on a 4-point scale from 0 (would never dose) to 3 (high change of dozing). The total score of the 8 items ranges from 0 to 24, with higher values indicating worse outcome. The overall number of baseline participants was based on the full analysis set (FAS)(n=44).
  units on a scale | 9.1 (4.7)
ISI total score [Mean (Standard Deviation); unit: units on a scale] — The Insomnia Severity Index (ISI) is a patient-rated scale desgined to measure the patient's perception of his/her insomnia. The ISI comprises 7 items.and each of the 7 items is rated on a 5-point scale from 0 (best situation) to 4 (worst situation). The total score of the 7 items ranges from 0 to 28, with higher values indicating worse outcome. The overall number of baseline participants was based on the full analysis set (FAS)(n=44).
  units on a scale | 19.4 (3.9)
CPFQ total score [Mean (Standard Deviation); unit: units on a scale] — The Cognitive and Physical Functioning Questionnaire (CPFQ) is a patient-rated scale designed to assess cognitive and executive dysfunction including symptoms of fatigue in mood and anxiety disorders. The CPFQ consists of 7 items, each rated on a scale from 1 (greater than normal functioning) to 6 (poorer than normal functioning). The total score of the 7 items ranges from 7 to 42, with higher values indicating worse outcome. The overall number of baseline participants was based on the full analysis set (FAS)(n=44).
  units on a scale | 27.1 (5.3)
BRIAN total score [Mean (Standard Deviation); unit: units on a scale] — The Biological Rhythms Interview of Assessment in Neuropsychiatry (BRIAN) is a clinician-rated scale designed to assess biological rhythms. The BRIAN consists of 18 items divided in 4 subscales: sleep (5 items), activity (5 items), social (4 items), and eating pattern (4 items). Each item is rated on a scale from 1 (no difficulties) to 4 (serious difficulties). The total score of the 18 items ranges from 18 to 72, with higher values indicating worse outcome. The overall number of baseline participants was based on the full analysis set (FAS)(n=44).
  units on a scale | 51.7 (10.3)

OUTCOME MEASURES:

1. Primary Outcome: Changes From Baseline to Week 8 on Sleep Quality as Assessed by Polysomnographic Recorded (PSG) Parameters
Description: The key PSG parameters assessed were the latency to persistent sleep (PSG LPS), sleep onset latency (PSG SOL), wake-time after sleep onset (PSG WASO), total sleep time (PSG TST), number of awakenings (PSG NAW), and sleep efficiency (PSG SE). The results for PSG LPS, PSG SOL, PSG WASO, and PSG TST are presented separately from the PSG NAW, and from the PSG SE due to the different units of measurement involved. As this was an open-label exploratory study, all outcomes should be considered as exploratory outcomes.
Time Frame: Baseline and Week 8
Population: The full-analysis set (FAS) comprised all patients treated, who had a valid baseline assessment and at least one valid post-baseline efficacy assessment. The analysis was performed using observed cases (OC) data.
Measure: Mean (Standard Error); unit: minutes (min)
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 44
minutes (min)
  PSG LPS (n=40) | -24.9 (4.8)
  PSG SOL (n=40) | -19.7 (3.8)
  PSG WASO (n=40) | -26.4 (6.1)
  PSG TST (n=41) | 49.0 (8.2)

2. Primary Outcome: Changes From Baseline to Week 8 on Sleep Quality as Assessed by Polysomnographic Recorded (PSG) Number of Awakenings (PSG NAW)
Description: as for outcome 1
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Mean (Standard Error); unit: number of events
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 40
number of events | 0.06 (0.8)

3. Primary Outcome: Changes From Baseline to Week 8 on Sleep Quality as Assessed by Polysomnographic Recorded (PSG) Sleep Efficiency (PSG SE)
Description: as for outcome 1
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Mean (Standard Error); unit: percentage (%)
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 41
percentage (%) | 10.4 (1.7)

4. Primary Outcome: Changes From Baseline to Week 8 on Sleep Quality as Assessed by the Consensus Sleep Diary for Morning (CSD-M) Sleep Efficiency (SE)
Description: The key CSD-M parameters assessed were the sleep efficiency (CSD-M SE), total sleep time (CSD-M TST), sleep onset latency (CSD-M SOL), wake-time after sleep onset (CSD-M WASO), and number of awakenings (CSD-M NAW). The results for CSD-M SE are presented separately from CSD-M TST, CSD-M SOL, and CSD-M WASO, and from CSD-M NAW due to the different units of measurement involved. As this was an open-label exploratory study, all outcomes should be considered as exploratory outcomes.
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Mean (Standard Error); unit: percentage of time
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 21
percentage of time | 13.4 (3.2)

5. Primary Outcome: Changes From Baseline to Week 8 on Sleep Quality as Assessed by the Consensus Sleep Diary for Morning (CSD-M)
Description: as for outcome 4
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Mean (Standard Error); unit: minutes (min)
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 44
minutes (min)
  CSD-M TST (n=21) | 69.9 (14.6)
  CSD-M SOL (n=21) | -37.1 (12.3)
  CSD-M WASO (n=21) | -42.9 (29.0)

6. Primary Outcome: Changes From Baseline to Week 8 on Sleep Quality as Assessed by the Consensus Sleep Diary for Morning (CSD-M) Number of Awakenings (NAW)
Description: The key CSD-M parameters assessed were the sleep efficiency (CSD-M SE), total sleep time (CSD-M TST), sleep onset latency (CSD-M SOL), wake-time after sleep onset (CSD-M WASO), and number of awakenings (CSD-M NAW). As this was an open-label exploratory study, all outcomes should be considered as exploratory outcomes.
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Mean (Standard Error); unit: number
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 21
number | 0.0 (0.5)

7. Primary Outcome: Changes From Baseline to Week 8 in Sleep Architecture as Assessed With Polysomnography
Description: The key sleep architecture parameters assessed with polysomnography were the percentage of time and duration spent in Stages N1 (non-rapid eye movement [non-REM]), N2 (non-REM), N3 (non-REM), and REM, respectively, as well as the duration of latency to REM sleep. The results for the percentage of time spent at each stage is presented separately from the duration due to the different units of measurement involved. As this was an open-label exploratory study, all outcomes should be considered as exploratory outcomes.
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Mean (Standard Error); unit: percentage of total sleep duration
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 44
percentage of total sleep duration
  Stage N1 (n=40) | -0.7 (0.7)
  Stage N2 (n=40) | 3.5 (1.5)
  Stage N3 (n=40) | -2.2 (0.8)
  Stage REM (n=40) | -0.6 (1.1)

8. Primary Outcome: Changes From Baseline to Week 8 in Sleep Architecture as Assessed With Polysomnography (Continued)
Description: as for outcome 7
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Mean (Standard Error); unit: minutes
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 44
minutes
  Stage N1 Duration (n=41) | 4.5 (2.5)
  Stage N2 Duration (n=41) | 43.1 (8.3)
  Stage N3 Duration (n=41) | -3.1 (3.0)
  Stage REM Duration (n=41) | 4.5 (4.4)
  Latency to REM Sleep Duration (n=38) | -16.2 (14.4)

9. Primary Outcome: Change From Baseline to Week 8 in ISI Total Score
Description: The Insomnia Severity Index (ISI) is a patient-rated scale desgined to measure the patient's perception of his/her insomnia. The ISI comprises 7 items: difficulty falling asleep, difficulty staying asleep, problems waking up early in the morning, satisfaction with current sleep pattern, interference with daily functioning, how much others notice the sleep problem impairs quality of life, and distress caused by the sleep problem. Each of the 7 items is rated on a 5-point scale from 0 (best situation) to 4 (worst situation). The total score of the 7 items ranges from 0 to 28, with higher values indicating worse outcome. As this was an open-label exploratory study, all outcomes should be considered as exploratory outcomes.
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 41
units on a scale | -9.2 (1.1)

10. Primary Outcome: Change From Baseline to Week 8 on ESS Total Score
Description: The Epworth Sleepiness Scale (ESS) is a is a patient-rated scale designed to measure daytime sleepiness. The ESS consists of 8 items describing different situations/activities and the patients rate the chance of them dozing off or falling asleep when they are in these situations. Each item is rated on a 4-point scale from 0 (would never dose) to 3 (high change of dozing). The total score of the 8 items ranges from 0 to 24, with higher values indicating worse outcome. As this was an open-label exploratory study, all outcomes should be considered as exploratory outcomes.
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 41
units on a scale | -2.6 (0.7)

11. Primary Outcome: Changes From Baseline to Week 8 in Response Speed as Assessed Using a PVT Device
Description: The psychomotor vigilance task (PVT) measures sustained or vigilant attention by recording response time (milliseconds) to a visual/or auditory stimulus that appears at random inter-stimulus intervals (range: from 2 to 10 seconds). The patient was instructed to monitor a red rectangular box on the computer screen and to press a response button as soon as a yellow stimulus counter appeared on the screen. The parameters assessed using a PVT device were response speed and number of lapses. The results for response speed is presented separately from the number of lapses due to the different units of measurement involved. As this was an open-label exploratory study, all outcomes should be considered as exploratory outcomes.
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Mean (Standard Error); unit: speed (per second)
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 40
speed (per second) | -0.2 (0.1)

12. Primary Outcome: Changes From Baseline to Week 8 in Number of Lapses as Assessed Using a PVT Device
Description: as for outcome 11
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Mean (Standard Error); unit: number
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 40
number | 2.1 (2.4)

13. Primary Outcome: Change From Baseline to Week 8 on BL-VAS-s (Evening) Score
Description: The Bond-Lader Visual Analogue Scale - Sedation (BL-VAS-s) is a patient-rated scale designed to assess the current level of sedation. The BL-VAS-s was assessed for the evening (19:00 to 23:59 hours), morning (00:00 to 08:59 hours) and at noon (11:00 to 13:59 hours). The BL-VAS-s is a single item scale rated on a 100mm visual analogue scale. The score is measured from the left to a mark made on the line by the patient and ranges from 0 (alert) to 100 (drowsy). As this was an open-label exploratory study, all outcomes should be considered as exploratory outcomes.
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 33
units on a scale | 1.4 (4.2)

14. Primary Outcome: Change From Baseline to Week 8 on BL-VAS-s (Morning) Score
Description: as for outcome 13
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 34
units on a scale | -9.2 (4.5)

15. Primary Outcome: Change From Baseline to Week 8 on BL-VAS-s Scores (Noon)
Description: as for outcome 13
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 23
units on a scale | -7.4 (6.7)

16. Primary Outcome: Change From Baseline to Week 8 in CPFQ Total Score
Description: The Cognitive and Physical Functioning Questionnaire (CPFQ) is a patient-rated scale designed to assess cognitive and executive dysfunction including symptoms of fatigue in mood and anxiety disorders. The CPFQ consists of 7 items, each rated on a scale from 1 (greater than normal functioning) to 6 (poorer than normal functioning). The total score of the 7 items ranges from 7 to 42, with higher values indicating worse outcome. As this was an open-label exploratory study, all outcomes should be considered as exploratory outcomes.
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 41
units on a scale | -8.4 (1.1)

17. Primary Outcome: Changes From Baseline to Week 8 in Circadian and Biological Rhythm
Description: The parameters used to assess circadian and biological rhythm were the time to peak cortisol concentration, time to dim-light melatonin onset (DLMO) and phase angle. As this was an open-label exploratory study, all outcomes should be considered as exploratory outcomes.
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Mean (Standard Error); unit: minutes
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 9
minutes
  Time to peak cortisol concentration | -60 (23)
  Time to DLMO | 48 (49)
  Phase angle | 108 (61)

18. Primary Outcome: Change From Baseline to Week 8 in MADRS Total Score
Description: The Montgomery Aasberg Depression Rating Scale (MADRS) is a 10-item rating scale designed to assess the severity of the symptoms in depressive illness and to be sensitive to treatment effects. Items in the scale assess apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, and suicidal thoughts. Symptoms are rated on a 7-point scale from 0 (no symptoms) to 6 (severe symptoms). Definitions of severity are provided at two-point intervals. The total score of the 10 items ranges from 0 to 60, with higher values indicating worse outcome. As this was an open-label exploratory study, all outcomes should be considered as exploratory outcomes.
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 41
units on a scale | -16.0 (1.7)

19. Primary Outcome: Change From Baseline to Week 8 in CGI-S Score
Description: The Clinical Global Impression - Severity of Illness (CGI-S) scale assesses the clinician's impression of the patient's current state of mental illness. The clinician uses his or her clinical experience of this patient population to rate the severity of the patient's current mental illness on a 7-point scale ranging from 1 (normal - not at all ill) to 7 (among the most extremely ill patients), with higher values indicating worse outcome. As this was an open-label exploratory study, all outcomes should be considered as exploratory outcomes.
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 41
units on a scale | -1.8 (0.2)

20. Primary Outcome: Percentage of MADRS Responders at Week 8
Description: The Montgomery Aasberg Depression Rating Scale (MADRS) is a 10-item rating scale designed to assess the severity of the symptoms in depressive illness and to be sensitive to treatment effects. Items in the scale assess apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, and suicidal thoughts. Symptoms are rated on a 7-point scale from 0 (no symptoms) to 6 (severe symptoms). Definitions of severity are provided at two-point intervals. The total score of the 10 items ranges from 0 to 60, with higher values indicating worse outcome. Response was defined as a ≥50% decrease in MADRS total score from baseline. As this was an open-label exploratory study, all outcomes should be considered as exploratory outcomes.
Time Frame: Week 8
Population: as for outcome 1
Measure: Number; unit: percentage of patients
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 41
percentage of patients | 56

21. Primary Outcome: Percentage of MADRS Remitters at Week 8
Description: The Montgomery Aasberg Depression Rating Scale (MADRS) is a 10-item rating scale designed to assess the severity of the symptoms in depressive illness and to be sensitive to treatment effects. Items in the scale assess apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, and suicidal thoughts. Symptoms are rated on a 7-point scale from 0 (no symptoms) to 6 (severe symptoms). Definitions of severity are provided at two-point intervals. The total score of the 10 items ranges from 0 to 60, with higher values indicating worse outcome. Remission was defined as a MADRS total score ≤10 and a ≥50% decrease in MADRS total score from baseline. As this was an open-label exploratory study, all outcomes should be considered as exploratory outcomes.
Time Frame: Week 8
Population: as for outcome 1
Measure: Number; unit: percentage of patients
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 41
percentage of patients | 54

22. Primary Outcome: Changes From Baseline to Week 8 on Sleep Quality as Assessed by Actigraphy (ACT) Parameters
Description: The key ACT parameters assessed were the total sleep time (ACT TST), wake-time after sleep onset (ACT WASO), sleep onset latency (ACT SOL), sleep efficiency (ACT SE), and the number of awakenings (ACT NAW). The results for ACT TST, ACT WASO, and ACT SOL are presented separately from ACT SE, and from ACT NAW, due to the different units of measurement involved. As this was an open-label exploratory study, all outcomes should be considered as exploratory outcomes.
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Mean (Standard Error); unit: minutes
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 44
minutes
  ACT TST (n=33) | -9.0 (15.7)
  ACT WASO (n=33) | -6.1 (6.5)
  ACT SOL (n=32) | -5.5 (3.6)

23. Primary Outcome: Changes From Baseline to Week 8 on Sleep Efficiency (SE) as Assessed by Actigraphy (ACT)
Description: The key ACT parameters assessed were the total sleep time (ACT TST), sleep efficiency (ACT SE), sleep onset latency (ACT SOL), wake-time after sleep onset (ACT WASO), and the number of awakenings (ACT NAW). The results for ACT TST, ACT SE, ACT WASO, and ACT NAW are presented separately from ACT SOL as the number of patients available for analysis was different. As this was an open-label exploratory study, all outcomes should be considered as exploratory outcomes.
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Mean (Standard Error); unit: percentage of time
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 33
percentage of time | -1.3 (3.7)

24. Primary Outcome: Changes From Baseline to Week 8 on Number of Awakenings (NAW) as Assessed by Actigraphy (ACT)
Description: as for outcome 23
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Mean (Standard Error); unit: number of events
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 33
number of events | -2.0 (1.1)

25. Primary Outcome: Change From Baseline to Week 8 in BRIAN Total Score
Description: The Biological Rhythms Interview of Assessment in Neuropsychiatry (BRIAN) is a clinician-rated scale designed to assess biological rhythms. The BRIAN consists of 18 items divided in 4 subscales: sleep (5 items), activity (5 items), social (4 items), and eating pattern (4 items). Each item is rated on a scale from 1 (no difficulties) to 4 (serious difficulties). The total score of the 18 items ranges from 18 to 72, with higher values indicating worse outcome. As this was an open-label exploratory study, all outcomes should be considered as exploratory outcomes.
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 41
units on a scale | -17.4 (1.9)

26. Primary Outcome: CGI-I Score at Week 8
Description: The Clinical Global Impression - Global Improvement (CGI-I) assesses the clinician's impression of the patient's improvement (or worsening). The clinician assesses the patient's condition relative to a baseline on a 7-point scale ranging from 1 (very much improved) to 7 (very much worse), with higher values indicating worse outcome. As this was an open-label exploratory study, all outcomes should be considered as exploratory outcomes.
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 41
units on a scale | 2.2 (1.1)

ADVERSE EVENTS:
Time Frame: Baseline to end of treatment (Week 8)
Groups:
- Brexpiprazole: The all-patients-treated set (APTS) comprises all patients who took at least one dose of brexpiprazole.
Arm/Group | Brexpiprazole
Serious Adverse Events (participants affected / at risk) | 0/44
Other Adverse Events (participants affected / at risk) | 22/44
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Brexpiprazole (N=44)
Nausea (Gastrointestinal disorders) | 6
Fatigue (General disorders) | 3
Upper respiratory tract infection (Infections and infestations) | 4
Weight increased (Investigations) | 4
Headache (Nervous system disorders) | 5
Sedation (Nervous system disorders) | 6
Somnolence (Nervous system disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No